CLINICAL TRIAL: NCT04652726
Title: Two Part (Double-blind Inclisiran Versus Placebo [Year 1] Followed by Open-label Inclisiran [Year 2]) Randomized Multicenter Study to Evaluate Safety, Tolerability, and Efficacy of Inclisiran in Adolescents (12 to Less Than 18 Years) With Heterozygous Familial Hypercholesterolemia and Elevated LDL-cholesterol (ORION-16)
Brief Title: Study to Evaluate Efficacy and Safety of Inclisiran in Adolescents With Heterozygous Familial Hypercholesterolemia
Acronym: ORION-16
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKJX839C12301; 2020-002757-18 (EudraCT Number)
Record Dates: First submitted 2020-12-02; First posted 2020-12-03 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Familial Hypercholesterolemia - Heterozygous
Keywords: Heterozygous familial hypercholesterolemia (HeFH); LDL-cholesterol (LDL-C); adolescents; pediatric; small interfering ribonucleic acid (siRNA)
MeSH Terms: interventions — ALN-PCS; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel (Year 1) to single-group (Year 2)
Who Masked: Participant, Investigator
Masking Description: Masked (Year 1) to No Masking (Year 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran (Experimental): Year 1 - inclisiran sodium 300 mg subcutaneous injection (given at Days 1, 90, and 270) Day 360 only - placebo subcutaneous injection Year 2 - inclisiran sodium 300 mg subcutaneous injection (given at Days 450 and 630)
  Interventions: Drug: Inclisiran
- Placebo (Placebo Comparator): Year 1 - placebo subcutaneous injection (given at Days 1, 90 and 270) Year 2 - inclisiran sodium 300 mg subcutaneous injection (given at Days 360, 450, and 630)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclisiran — Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) in 1.5 mL solution for subcutaneous injection
  Other Names: KJX839
  Arms: Inclisiran
Drug: Placebo — Sterile normal saline (0.9% sodium chloride in water for subcutaneous injection)
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
This was a pivotal phase III study designed to evaluate safety, tolerability, and efficacy of inclisiran in adolescents with heterozygous familial hypercholesterolemia (HeFH) and elevated low density lipoprotein cholesterol (LDL-C).

DETAILED DESCRIPTION:
This was a two-part (1 year double-blind inclisiran versus placebo / 1 year open-label inclisiran) multicenter study designed to evaluate safety, tolerability, and efficacy of inclisiran in adolescents with heterozygous familial hypercholesterolemia (HeFH) and elevated low density lipoprotein cholesterol (LDL-C) on stable standard of care background lipid-lowering therapy. The primary objective was to demonstrate superiority of inclisiran compared to placebo in reducing LDL-C (percent change) at Day 330.

ELIGIBILITY:
Inclusion Criteria:

* Heterozygous Familial Hypercholesterolemia (HeFH) diagnosed either by genetic testing or on phenotypic criteria
* Fasting LDL-C >130 mg/dL (3.4 mmol/L) at screening
* Fasting triglycerides <400 mg/dL (4.5 mmol/L) at screening
* On maximally tolerated dose of statin (investigator's discretion) with or without other lipid-lowering therapy; stable for ≥ 30 days before screening

Exclusion Criteria:

* Homozygous familial hypercholesterolemia (HoFH)
* Active liver disease
* Secondary hypercholesterolemia, e.g. hypothyroidism or nephrotic syndrome
* Previous treatment with monoclonal antibodies directed towards PCSK9 (within 90 days of screening)
* Recent and/or planned use of other investigational medicinal products or devices

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (57):
- United States (6):
  - Tucson Medical Center, Tucson, Arizona
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Wake Forest U of Health Sciences, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Childrens Hospital Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Primary Children's Medical Center, Salt Lake City, Utah
- Novartis Investigative Site, Formosa, Formosa Province, Argentina
- Brazil (4):
  - Unidade de pesquisa clinica - Hospital Universitario Walter Cantidio, Fortaleza, Ceará
  - Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Setor de Lípides, Aterosclerose e Biologia, São Paulo, São Paulo
  - Heart Institute (InCOr) HCMFUSP, São Paulo, São Paulo
- Novartis Investigative Site, Québec, Quebec, Canada
- Novartis Investigative Site, Prague, Czechia
- France (3):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Toulouse
- Germany (3):
  - Universitaetsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - KKIM UK Frankfurt/Main, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- Greece (3):
  - University General Hospital of Ioannina, Ioannina, GR
  - Hippokrateion General Hospital of Athens Greece, Athens
  - Metropolitan Hospital, Athens
- Novartis Investigative Site, Pécs, Hungary
- Israel (2):
  - Lipid Research, Jerusalem
  - Lipids Center Sheba Medical Center, Israel, Ramat Gan
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Irbid, Jordan
- Hotel Dieu de France Hospital, El Achrafiyé, Lebanon
- UiTM Sungai Buloh, Sungai Buloh, Selangor, Malaysia
- Netherlands (2):
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Amsterdam
- Novartis Investigative Site, Oslo, Norway
- Poland (2):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz
- Russia (3):
  - Institute of the complex problems of cardiovascular disease, Kemerovo
  - Novartis Investigative Site, Moscow
  - Institute of Internal Prev. Med., Novosibirsk
- Novartis Investigative Site, Poprad, Slovakia
- University Medical Centre Ljubljana, Div. of Pediatric Dept. of Endocrinology, Diabetes and Metabolic Diseases, Ljubljana, Slovenia
- South Africa (3):
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Somerset West, Western Cape
  - Novartis Investigative Site, Cape Town
- Spain (5):
  - Hospital Reina Sofia, Córdoba, Andalusia
  - Hospital Virgen de la Vcitoria, Málaga, Andalusia
  - Novartis Investigative Site, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Abente y Lago, A Coruña
- Novartis Investigative Site, Geneva, Switzerland
- Taiwan (2):
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Adana
  - Gazi University Medical Faculty, Ankara
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Wiegman A, Peterson AL, Bruckert E, Defesche JC, Schweizer A, Bergeron J, Chueca MJ, Roeters van Lennep JE, Santos RD, Schwab KO, Lesogor A, Zhang S, Hegele RA. Efficacy and safety of inclisiran in adolescents with heterozygous familial hypercholesterolaemia (ORION-16): a two-part, randomised, multicentre clinical trial. Lancet Diabetes Endocrinol. 2026 Jan 27:S2213-8587(25)00351-1. doi: 10.1016/S2213-8587(25)00351-1. Online ahead of print. PMID 41616799
- [Derived] Reijman MD, Schweizer A, Peterson ALH, Bruckert E, Stratz C, Defesche JC, Hegele RA, Wiegman A. Rationale and design of two trials assessing the efficacy, safety, and tolerability of inclisiran in adolescents with homozygous and heterozygous familial hypercholesterolaemia. Eur J Prev Cardiol. 2022 Jul 20;29(9):1361-1368. doi: 10.1093/eurjpc/zwac025. PMID 35175352
- [Derived] Warden BA, Duell PB. Inclisiran: A Novel Agent for Lowering Apolipoprotein B-containing Lipoproteins. J Cardiovasc Pharmacol. 2021 Aug 1;78(2):e157-e174. doi: 10.1097/FJC.0000000000001053. PMID 33990512
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2617
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 141 participants were randomized in 26 countries and 51 study centers:Argentina (1), Brazil (3), Canada (1), Czech Republic (2), France (3), Germany (2), Greece (1), Hungary (1), Israel (2), Italy (4), Jordan (1), Lebanon (1), Malaysia (1), Netherlands (2), Norway (1), Poland (2), Russian Federation (2), Slovakia (1), Slovenia (1), South Africa (3), Spain (4), Switzerland (1), Taiwan (1), Turkey (4), United Kingdom (1), and United States of America (5).
Pre-assignment Details: The study had an approximately 4-week screening/run-in period
Groups:
- Part 1- Inclisiran: Inclisiran sodium 300 mg subcutaneous (sc) injection (given at Days 1, 90 and 270)
- Part 1 - Placebo: Placebo sc injection (given at Day 1, 90 and 270)
- Part 2 - Inclisiran (Total): Inclisiran sodium 300 mg sc injection (given at Days 450 and 630). In addition, participants assigned to placebo in Part 1 received inclisiran sodium 300 mg sc injection on Day 360, while participants assigned to inclisiran in Part 1 received placebo sc injection on Day 360
Period: Part 1 (Double-blind Period)
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Started | 93 | 48 | 0
Completed | 91 | 48 | 0
Not Completed | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Participant/guardian decision | 1 | 0 | 0
Period: Part 2 (Open-label Period)
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Started | 0 | 0 | 139
Completed | 0 | 0 | 139
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics are based on all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Total
Number analyzed (Participants) | 93 | 48 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 93 | 48 | 141
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (2.02) | 14.9 (1.80) | 15.1 (1.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 24 | 75
  Male | 42 | 24 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 0 | 4
  Black or African American | 5 | 0 | 5
  Other | 4 | 0 | 4
  White | 80 | 48 | 128

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in LDL-C From Baseline to Day 330 (Part 1/Year 1)
Description: Percentage change in low-density lipoprotein cholesterol (LDL-C) from baseline to Day 330 (Year 1)
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change in LDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 93 | 48
percent change in LDL-C | -27.14 [-32.04 to -22.24] | 1.40 [-3.97 to 6.78]
Statistical Analysis 1: Comparison: Part 1- Inclisiran vs Part 1 - Placebo; Test type: Superiority; p < .0001, ANCOVA; LS Mean = -28.54, 95% CI 2-sided [-35.81 to -21.27]

2. Secondary Outcome: Time-adjusted Percent Change in LDL-C From Baseline After Day 90 and up to Day 330 (Part 1/Year 1)
Description: Time-adjusted percent change in LDL-C (after Day 90 and up to Day 330), calculated as the average of percent changes from baseline to Days 150, 270 and 330
Time Frame: Baseline, after Day 90 up to Day 330
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: Time-adjusted percent change in LDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 93 | 48
Time-adjusted percent change in LDL-C | -26.04 [-30.11 to -21.98] | 3.26 [-2.37 to 8.89]
Statistical Analysis 1: Comparison: Part 1- Inclisiran vs Part 1 - Placebo; Test type: Superiority; p < .0001, MMRM; LS Mean = -29.30, 95% CI 2-sided [-36.24 to -22.36]

3. Secondary Outcome: Absolute Change in LDL-C From Baseline to up Day 330 (Part 1/Year 1)
Description: Absolute change in LDL-C from baseline to Day 330.
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 93 | 48
mg/dL | -50.54 [-59.22 to -41.86] | -0.55 [-10.48 to 9.38]
Statistical Analysis 1: Comparison: Part 1- Inclisiran vs Part 1 - Placebo; Test type: Superiority; p < .0001, ANCOVA; LS Mean = -49.99, 95% CI 2-sided [-63.18 to -36.81]

4. Secondary Outcome: Percent Change in Apo B From Baseline up to Day 330 (Part 1/Year 1)
Description: Percentage change in apolipoprotein B (Apo B) from baseline to Day 330.
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change in Apo B
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 93 | 48
Percent change in Apo B | -21.46 [-25.59 to -17.33] | 4.24 [-0.07 to 8.56]
Statistical Analysis 1: Comparison: Part 1- Inclisiran vs Part 1 - Placebo; Test type: Superiority; p < .0001, ANCOVA; LS Mean = -25.70, 95% CI 2-sided [-31.68 to -19.73]

5. Secondary Outcome: Percent Change in Lp(a) From Baseline up to Day 330 (Part 1/Year 1)
Description: Percentage change in lipoprotein (a) [Lp(a)] from baseline to Day 330.
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change in Lp(a)
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 93 | 48
Percent change in Lp(a) | -5.04 [-14.21 to 4.13] | 1.14 [-5.48 to 7.77]
Statistical Analysis 1: Comparison: Part 1- Inclisiran vs Part 1 - Placebo; Test type: Superiority; p = 0.1419, ANCOVA; LS Mean = -6.18, 95% CI 2-sided [-17.48 to 5.12]

6. Secondary Outcome: Percent Change in Non-HDL-C From Baseline up to Day 330 (Part 1/Year 1)
Description: Percentage change in non-high density lipoprotein cholesterol (non-HDL-C) from baseline to Day 330.
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change in non-HDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 93 | 48
Percent change in non-HDL-C | -25.04 [-29.68 to -20.41] | 1.76 [-3.25 to 6.77]
Statistical Analysis 1: Comparison: Part 1- Inclisiran vs Part 1 - Placebo; Test type: Superiority; p < .0001, ANCOVA; LS Mean = -26.80, 95% CI 2-sided [-33.63 to -19.97]

7. Secondary Outcome: Percent Change in Total Cholesterol From Baseline up to Day 330 (Part 1/Year 1)
Description: Percentage change in total cholesterol from baseline to Day 330.
Time Frame: Baseline and Day 330
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change in total cholesterol
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 93 | 48
Percent change in total cholesterol | -18.72 [-22.48 to -14.96] | 0.48 [-3.46 to 4.42]
Statistical Analysis 1: Comparison: Part 1- Inclisiran vs Part 1 - Placebo; Test type: Superiority; p < .0001, ANCOVA; LS Mean = -19.20, 95% CI 2-sided [-24.65 to -13.75]

8. Secondary Outcome: Percent Change in LDL-C From Baseline up to Day 720
Description: Percentage change in LDL-C from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned by randomization. At each time point, only subjects with a value at both baseline and that time point are included.
Measure: Mean (Standard Deviation); unit: Percent change in LDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 93 | 48 | 139
Percent change in LDL-C
  DAY 90: number analyzed (Participants) | 93 | 48 | 0
  DAY 90 | -23.9 (22.14) | -0.1 (20.16) |
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | -32.5 (21.47) | 6.4 (28.83) |
  DAY 270: number analyzed (Participants) | 92 | 48 | 0
  DAY 270 | -19.0 (28.31) | 2.1 (22.44) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -27.8 (22.95) | 1.5 (20.59) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -26.1 (22.71) | 1.5 (30.56) |
  DAY 450: number analyzed (Participants) | 0 | 0 | 139
  DAY 450 |  |  | -24.5 (26.45)
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | -32.5 (22.80)
  DAY 630: number analyzed (Participants) | 0 | 0 | 139
  DAY 630 |  |  | -26.5 (24.33)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -33.7 (23.98)

9. Secondary Outcome: Absolute Change in LDL-C From Baseline up to Day 720
Description: Absolute change in LDL-C from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 93 | 48 | 139
mg/dL
  DAY 90: number analyzed (Participants) | 93 | 48 | 0
  DAY 90 | -45.4 (45.26) | -3.0 (35.02) |
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | -61.0 (45.84) | 6.6 (46.22) |
  DAY 270: number analyzed (Participants) | 92 | 48 | 0
  DAY 270 | -38.4 (55.77) | 1.0 (36.92) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -51.9 (45.47) | -0.3 (38.04) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -49.0 (44.49) | -2.9 (51.74) |
  DAY 450: number analyzed (Participants) | 0 | 0 | 139
  DAY 450 |  |  | -46.3 (52.51)
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | -60.8 (48.88)
  DAY 630: number analyzed (Participants) | 0 | 0 | 139
  DAY 630 |  |  | -50.9 (50.30)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -64.1 (53.91)

10. Secondary Outcome: Percent Change in Apo B From Baseline up to Day 720
Description: Percentage change in apolipoprotein B (Apo B) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change in Apo B
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
Percent change in Apo B
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | -25.1 (18.18) | 2.2 (20.77) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -21.9 (19.51) | 3.9 (18.13) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -19.3 (21.36) | 1.7 (22.70) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 138
  DAY 510 |  |  | -24.5 (21.77)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -25.7 (21.71)

11. Secondary Outcome: Absolute Change in Apo B From Baseline up to Day 720
Description: Absolute change in apolipoprotein B (Apo B) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
mg/dL
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | -33.3 (28.20) | 0.0 (27.38) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -29.2 (28.04) | 2.9 (23.47) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -26.1 (29.59) | -0.6 (28.72) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 138
  DAY 510 |  |  | -33.5 (32.13)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -35.4 (33.83)

12. Secondary Outcome: Percent Change in Lp(a) From Baseline up to Day 720
Description: Percentage change in lipoprotein (a) [Lp(a)] from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change in Lp(a)
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
Percent change in Lp(a)
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | -13.4 (22.60) | 5.4 (23.96) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -7.2 (30.80) | 1.1 (24.25) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -9.3 (28.44) | 3.6 (23.27) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | -13.3 (28.81)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -4.2 (163.74)

13. Secondary Outcome: Absolute Change in Lp(a) From Baseline up to Day 720
Description: Absolute change in lipoprotein (a) [Lp(a)] from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
nmol/L
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | -12.5 (34.73) | 3.2 (20.67) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -9.5 (33.81) | 5.3 (21.55) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -10.2 (31.16) | 4.4 (22.99) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | -10.1 (34.98)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -9.0 (50.08)

14. Secondary Outcome: Percent Change in Non-HDL-C From Baseline up to Day 720
Description: Percentage change in non-high density lipoprotein cholesterol (non-HDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change in non-HDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
Percent change in non-HDL-C
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | -29.0 (20.15) | 5.1 (24.85) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -25.7 (21.69) | 1.8 (19.43) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -24.0 (21.74) | 1.2 (27.43) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | -29.9 (21.60)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -31.0 (23.04)

15. Secondary Outcome: Absolute Change in Non-HDL-C From Baseline up to Day 720
Description: Absolute change in non-high density lipoprotein cholesterol (non-HDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
mg/dL
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | -60.2 (47.41) | 5.7 (47.61) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -52.6 (46.93) | 0.5 (39.20) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -49.7 (46.30) | -3.0 (52.75) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | -62.0 (51.09)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -65.1 (56.16)

16. Secondary Outcome: Percent Change in Total Cholesterol From Baseline up to Day 720
Description: Percentage change in total cholesterol from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change in total cholesterol
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
Percent change in total cholesterol
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | -22.6 (15.77) | 4.4 (20.49) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -19.2 (17.77) | 0.6 (15.46) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -18.5 (17.18) | 0.6 (21.81) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | -23.0 (17.50)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -23.7 (18.29)

17. Secondary Outcome: Absolute Change in Total Cholesterol From Baseline up to Day 720
Description: Absolute change in total cholesterol from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
mg/dL
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | -59.0 (47.79) | 6.6 (48.08) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -49.4 (47.77) | -0.9 (38.48) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -48.2 (47.06) | -3.1 (52.66) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | -59.6 (51.06)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -62.3 (55.05)

18. Secondary Outcome: Percent Change in Triglycerides From Baseline up to Day 720
Description: Percentage change in triglycerides from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change in triglycerides
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
Percent change in triglycerides
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | 16.2 (78.18) | 2.8 (37.44) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | 1.8 (38.39) | 9.7 (43.04) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | 1.7 (40.03) | 3.8 (35.76) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | 3.4 (43.08)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | 1.9 (41.84)

19. Secondary Outcome: Absolute Change in Triglycerides From Baseline up to Day 720
Description: Absolute change in triglycerides from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
mg/dL
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | 6.9 (64.67) | -4.8 (31.53) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -2.9 (35.01) | 3.5 (35.55) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -3.1 (38.13) | -1.7 (28.47) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | -4.2 (34.70)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -4.8 (36.21)

20. Secondary Outcome: Percent Change in HDL-C From Baseline up to Day 720
Description: Percentage change in high density lipoprotein cholesterol (HDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change in HDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
Percent change in HDL-C
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | 3.6 (18.88) | 3.6 (16.49) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | 7.4 (19.15) | -1.9 (16.15) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | 4.4 (19.54) | 0.9 (12.39) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | 6.6 (19.84)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | 7.4 (20.40)

21. Secondary Outcome: Absolute Change in HDL-C From Baseline up to Day 720
Description: Absolute change in high density lipoprotein cholesterol (HDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
mg/dL
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | 1.2 (10.23) | 0.9 (8.07) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | 3.2 (9.57) | -1.4 (7.77) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | 1.5 (9.59) | -0.1 (6.23) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | 2.4 (9.32)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | 2.8 (9.75)

22. Secondary Outcome: Percent Change in VLDL-C From Baseline up to Day 720
Description: Percentage change in very low density lipoprotein cholesterol (VLDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change in VLDL-C
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
Percent change in VLDL-C
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | 11.8 (60.04) | 3.3 (38.25) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | 0.6 (39.00) | 10.0 (42.29) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | 1.0 (40.15) | 4.7 (35.65) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | 1.4 (41.13)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | 1.9 (42.20)

23. Secondary Outcome: Absolut Change in VLDL-C From Baseline up to Day 720
Description: Absolute change in very low density lipoprotein cholesterol (VLDL-C) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
mg/dL
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | 0.7 (10.02) | -0.9 (6.37) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | -0.7 (7.04) | 0.8 (7.07) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | -0.7 (7.63) | -0.2 (5.66) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 139
  DAY 510 |  |  | -1.2 (6.90)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | -1.0 (7.40)

24. Secondary Outcome: Percent Change in Apo A1 From Baseline up to Day 720
Description: Percentage change in apolipoprotein A1 (Apo A1) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change in Apo A1
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
Percent change in Apo A1
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | 3.7 (15.40) | 0.4 (13.22) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | 5.2 (14.49) | -1.5 (10.58) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | 3.0 (15.12) | -1.5 (9.98) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 138
  DAY 510 |  |  | 6.3 (16.19)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | 4.9 (15.56)

25. Secondary Outcome: Absolute Change in Apo A1 From Baseline up to Day 720
Description: Absolute change in apolipoprotein A1 (Apo A1) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 92 | 48 | 139
mg/dL
  DAY 150: number analyzed (Participants) | 92 | 48 | 0
  DAY 150 | 3.3 (21.76) | 0.0 (17.72) |
  DAY 330: number analyzed (Participants) | 90 | 48 | 0
  DAY 330 | 6.1 (21.16) | -2.8 (14.24) |
  DAY 360: number analyzed (Participants) | 90 | 48 | 0
  DAY 360 | 2.7 (21.87) | -2.6 (13.89) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 138
  DAY 510 |  |  | 7.5 (22.24)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 139
  Day 720 (study completion) |  |  | 5.4 (21.61)

26. Secondary Outcome: Percent Change in PCSK9 From Baseline up to Day 720
Description: Percentage change in proprotein convertase subtilisin/kexin type 9 (PCSK9) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change in PCSK9
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 90 | 48 | 136
Percent change in PCSK9
  DAY 90: number analyzed (Participants) | 89 | 47 | 0
  DAY 90 | -67.8 (15.17) | 11.6 (46.61) |
  DAY 150: number analyzed (Participants) | 90 | 47 | 0
  DAY 150 | -72.3 (11.37) | 3.8 (36.95) |
  DAY 330: number analyzed (Participants) | 89 | 47 | 0
  DAY 330 | -72.9 (12.12) | 4.8 (34.50) |
  DAY 360: number analyzed (Participants) | 89 | 48 | 0
  DAY 360 | -72.0 (10.47) | 11.7 (57.77) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 136
  DAY 510 |  |  | -74.3 (10.46)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 136
  Day 720 (study completion) |  |  | -71.6 (13.42)

27. Secondary Outcome: Absolut Change in PCSK9 From Baseline up to Day 720
Description: Absolute change in proprotein convertase subtilisin/kexin type 9 (PCSK9) from baseline to each assessment time up to Day 720.
Time Frame: Baseline, up to Day 720
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1- Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
Number analyzed (Participants) | 90 | 48 | 136
ng/mL
  DAY 90: number analyzed (Participants) | 89 | 47 | 0
  DAY 90 | -259.6 (121.5) | 2.1 (223.16) |
  DAY 150: number analyzed (Participants) | 90 | 47 | 0
  DAY 150 | -274.8 (116.2) | -27.7 (210.44) |
  DAY 330: number analyzed (Participants) | 89 | 47 | 0
  DAY 330 | -278.2 (119.8) | -23.9 (210.85) |
  DAY 360: number analyzed (Participants) | 89 | 48 | 0
  DAY 360 | -275.4 (117.2) | -9.1 (245.36) |
  DAY 510: number analyzed (Participants) | 0 | 0 | 136
  DAY 510 |  |  | -288.1 (156.9)
  Day 720 (study completion): number analyzed (Participants) | 0 | 0 | 136
  Day 720 (study completion) |  |  | -279.5 (159.2)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 90 days post treatment or 30 days after last study visit, whichever was longer, up to a maximum duration of approximately 2 years.
Groups:
- Part 1 - Inclisiran: Inclisiran sodium 300 mg subcutaneous (sc) injection (given at Days 1, 90 and 270)
Arm/Group | Part 1 - Inclisiran | Part 1 - Placebo | Part 2 - Inclisiran (Total)
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/48 | 0/139
Serious Adverse Events (participants affected / at risk) | 3/93 | 1/48 | 6/139
Other Adverse Events (participants affected / at risk) | 57/93 | 29/48 | 52/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Inclisiran (N=93) | Part 1 - Placebo (N=48) | Part 2 - Inclisiran (Total) (N=139)
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Status migrainosus (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Inclisiran (N=93) | Part 1 - Placebo (N=48) | Part 2 - Inclisiran (Total) (N=139)
Nausea (Gastrointestinal disorders) | 4 | 1 | 4
Vomiting (Gastrointestinal disorders) | 5 | 1 | 0
Fatigue (General disorders) | 4 | 1 | 0
Influenza like illness (General disorders) | 4 | 3 | 2
Injection site pain (General disorders) | 4 | 2 | 4
Injection site reaction (General disorders) | 8 | 1 | 5
Malaise (General disorders) | 0 | 2 | 0
COVID-19 (Infections and infestations) | 17 | 12 | 7
Gastroenteritis (Infections and infestations) | 4 | 1 | 3
Influenza (Infections and infestations) | 10 | 6 | 11
Nasopharyngitis (Infections and infestations) | 13 | 9 | 14
Pharyngitis (Infections and infestations) | 4 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 2 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 1 | 1
Headache (Nervous system disorders) | 12 | 3 | 6
Migraine (Nervous system disorders) | 4 | 0 | 2
Syncope (Nervous system disorders) | 5 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT04652726/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT04652726/SAP_001.pdf